CLINICAL TRIAL: NCT01201109
Title: Five Years Follow-up After Carpal Tunnel Release in Diabetic and Non-diabetic Patients
Brief Title: Carpal Tunnel Release in Diabetic Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Skane University Hospital (Other)
Responsible Party: Niels Thomsen, MD, PhD, Dept of Hand Surgery, Skåne University Hospital, Malmö
Other Study IDs: 2010/354
Record Dates: First submitted 2010-09-13; First posted 2010-09-14 (Estimated); Last update posted 2010-09-28 (Estimated); Status verified 2010-09

CONDITIONS: Carpal Tunnel Syndrome; Diabetes; Nerve Entrapment
Keywords: Carpal tunnel syndrome; Entrapment neuropathies; Diabetes
MeSH Terms: conditions — Carpal Tunnel Syndrome; Diabetes Mellitus; Nerve Compression Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Diabetics: Diabetic patients operated for carpal tunnel syndrome
- Non-diabetics: Non-diabetic patients operated for carpal tunnel syndrome

SUMMARY:
The aim of this study is to extend a previously reported 1 year follow-up on carpal tunnel release, in matched diabetic and non-diabetic patients,to compare outcomes 5 years after surgery.

DETAILED DESCRIPTION:
The Follow-up investigation includes:

1. Clinical examination of sensory and motor function
2. Generic and disease specific self-administered questionnaires
3. Nerve conduction study
4. Vibration threshold testing

ELIGIBILITY:
Inclusion Criteria:

* diabetic and non-diabetic patients operated for carpal tunnel syndrome 5 years ago.

Exclusion Criteria:

* previous carpal tunnel release in the hand under study
* clinical signs of nerve entrapment other than CTS
* cervical radiculopathy, inflammatory joint disease
* renal failure
* thyroid disorders
* previous wrist fracture on the affected side
* daily long-term exposure to vibrating tools
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective series of matched diabetic and non-diabetic patients who were operated for carapl tunnel syndrome 5 years ago.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2010-11; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Patient self-reported outcome questionnaire | 5 years after carpal tunnel release
  Measured by 1). Boston Carpal Tunnel Questionnaire regarding carpal tunnel symptoms and disability. 2). Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36) registering health-related quality of life. 3). Cold intolerance on a CISS score

SECONDARY OUTCOMES:
Nerve conduction study and vibrotactile sense | 5 years after carpal tunnels release
  Change in Median nerve function by measuring Distal motor latency and antidromic sensory conduction velocity over the carpal tunnel segment.
  Evaluate development of peripheral neuropathy by measure of sural nerve sensory conduction velocity, sural nerve amplitude and peroneal nerve motor conduction velocity.
  Vibrotactile sense of the hand measured at 7 difference frequences from 5 - 500 Hz.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Dahlin, Md, PhD, Study Chair
Locations (1):
- Dept of Hand Surgery, Skåne University Hospital, Malmo, Sweden

REFERENCES:
- [Derived] Thomsen NOB, Dahlin LB. Vibrotactile sense 5 years after carpal tunnel release in people with diabetes: A prospective study with matched controls. Diabet Med. 2021 Jul;38(7):e14453. doi: 10.1111/dme.14453. Epub 2020 Nov 26. PMID 33169372